CLINICAL TRIAL: NCT04047017
Title: Camrelizumab Combined With Apatinib for Recurrent Resistant Gestational Trophoblastic Neoplasia: a Phase 2, Single-arm, Prospective Study
Brief Title: Camrelizumab Combined With Apatinib for Recurrent Resistant GTN
Acronym: GTN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, xiang yang, Chief, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-GTN-MUL-IIT-SHR1210-APA
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Gestational Trophoblastic Disease
Keywords: camrelizumab; apatinib; gestational trophoblastic neoplasia; high-risk; chemo-refractory; relapse
MeSH Terms: conditions — Gestational Trophoblastic Disease; Recurrence | interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Camrelizumab(SHR-1210) 200mg, once every 2 weeks, each 4 weeks is 1cycle. Apatinib :250 mg po qd
  Interventions: Drug: Apatinib; Drug: Camrelizumab

INTERVENTIONS:
Drug: Apatinib — 250mg, po, qd
Drug: Camrelizumab — 200mg, q2w

SUMMARY:
This study is to evaluate the efficacy and safety of camrelizumab plus apatinib in patients with high-risk chemo-refractory or relapsed GTN.

DETAILED DESCRIPTION:
Apatinib is an oral small-molecule tyrosine kinase inhibitor that selectively binds to and inhibits VEGF receptor 2. Novel immunotherapy using the immune checkpoint inhibitors such as anti-PD-1 antibody has received much attention. Camrelizumab as one of the anti-PD-1 drug have impressive clinical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent resistant GTN previously received twice or more combination chemotherapy before enrolment;
2. In the 20000 FIGO staging and classification, a risk score of 7 and above 7 (Considered high risk) or resistant recurrent placental site trophoblastic tumor or resistant recurrent epithelial trophoblastic tumor;
3. Aged 18-70 years;
4. An Eastern Cooperative Oncology Group performance status of 0-2;
5. abnormal serum HCG level;
6. Expected survival ≥ 4 months;
7. The function of vital organs meets the following requirements： Hemoglobin≥80g/L; Absolute neutrophil count≥1.5*109/L；Platelets≥100

   *109/L; Creatinine≤1.5 times ULN; Urea nitrogen≤2.5 times ULN; Total Bilirubin≤ULN; ALT and AST ≤ 2.5 times ULN; Albumin≥25g/L; TSH≤ULN(if TSH is abnormal, normal T3 and T4 also can acceptable)
8. Female subjects of childbearing age must exclude pregnancy and are willing to use a medically approved high-efficiency contraceptive (eg, IUD, contraceptive or condom) during the study period and within 3 months of the last study drug administration.
9. The subject should be aware of the purpose of the study and the operations required by the study and volunteer to participate in the study before sign the informed consent form

Exclusion Criteria:

1. Previously exposed to other anti-angiogenic small-molecule TKI drugs, such as pazopanib, sorafenib, regorafenib, cilnitraz, etc. or anti-angiogenic mAbs such as bevacizumab ; or had used an anti-PD-1 antibody, an anti-CTLA-4 antibody, TCR-T, CAR-T and other immune therapy; or 4 weeks before the first administration participated in any other clinical trials of anticancer drugs; or before the first dose Live attenuated vaccines are accepted within 4 weeks or during the study period.
2. Other malignant tumors have occurred in the past 3 years..
3. Immunosuppressive drugs used within 14 days prior to the first use of SHR-1210, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (ie, no more than 10 mg/day of turmeric or equivalent drug physiological dose) Other corticosteroids).
4. Late-stage patients with symptomatic, disseminated to visceral, short-term risk of life-threatening complications (including uncontrolled large amounts of exudate [thoracic, pericardium, abdominal cavity], pulmonary lymphangitis, and more than 30% liver involvement patients).
5. Any active autoimmune diseases or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, decreased thyroid function; subjects with vitiligo or complete remission asthma in childhood and without any intervention, all above can be included; asthma requiring medical intervention for bronchodilators should be excluded).
6. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite with the optimal medical treatment.
7. Grade II or higher myocardial ischemia, myocardial infarction or poor control arrhythmia (including male with QTc interval ≥ 450ms, or female with QTc interval≥ 470ms). According to NYHA criteria, grade III to IV cardiac insufficiency, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%; myocardial infarction occurred within 6 months before enrollment, New York Heart Association Level II or above failure, uncontrolled angina, uncontrolled severe ventricular arrhythmia, pericardial disease with clinically significant, or electrocardiogram suggesting acute ischemia or abnormal active conduction system.
8. Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5ULN), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy.
9. Half of a teaspoons (2.5 ml) or more hemoptysis was found within the first 2 months or there were significant clinical bleeding symptoms or clearly propensity bleeding within 3 months before participant in the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ or above in baseline or vasculitis; artery or venous thrombosis events within 6 months prior to the study, such as cerebrovascular accidents (Including transient ischemic attacks, cerebral hemorrhage, cerebral infarction, deep vein thrombosis and pulmonary embolism.
10. Severe infections within 4 weeks prior to accept medication (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever during screening/first administration >38.5 °C
11. Those who have a history of psychotropic drug abuse and are unable to quit or have mental disorders.
12. Major surgical procedures were performed within 4 weeks before the first administration. Or open wounds or fractures.
13. There are obvious factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction. Or sinus or perforation of empty organs within 6 months.
14. Routine urine test indicated that urinary protein (++) or more, confirmed urinary protein (>1.0 g) within 24 hours.
15. Patients with a history of allergy may be potentially allergic or intolerant to Apatinib and biological agents SHR-1210.
16. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA (> 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of the analysis method) or co-infection with hepatitis B and hepatitis C.
17. There is any situation that may damage the subject or cause the subject to fail to meet or implement the research requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
ORR(objective response rate) | Up to one years
  the proportion of patients with complete or partial response according to serum hCG level

SECONDARY OUTCOMES:
DoR（duration of response） | Up to one years
  time from the first evidence of response to disease progression or death, whichever came first
PFS(progression free survival) | Up to one years
  time from the treatment initiation to disease progression according to serum hCG level or death, whichever came first
OS (overall survival) | Up to one years
  time from the treatment initiation to the date of death or end of follow-up
Safety as measured by adverse events | Up to one years
  A NCI-CTC AE5.0 version was used to evaluate the grade of adverse reactions of the drug, to observe any adverse events and serious adverse events that occurred in all subjects during the clinical study period, including abnormal laboratory examination value, clinical manifestation symptoms and vital signs, to record their clinical manifestation characteristics, severity, occurrence time, duration, treatment method and prognosis, and to determine their correlation with the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng H, Zong L, Kong Y, Wang X, Gu Y, Cang W, Zhao J, Wan X, Yang J, Xiang Y. Camrelizumab plus apatinib in patients with high-risk chemorefractory or relapsed gestational trophoblastic neoplasia (CAP 01): a single-arm, open-label, phase 2 trial. Lancet Oncol. 2021 Nov;22(11):1609-1617. doi: 10.1016/S1470-2045(21)00460-5. Epub 2021 Oct 5. PMID 34624252